CLINICAL TRIAL: NCT04370340
Title: Application of a Perineal Protection Device in Vacuum-assisted Births: a Prospective Randomized Controlled Trial
Brief Title: Application of a Perineal Protection Device in Vacuum-assisted Births
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PeriProtectTrial
Record Dates: First submitted 2020-04-21; First posted 2020-04-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Vaginal Tear; Perineal Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- intervention (Active Comparator)
  Interventions: Device: BabySlide

INTERVENTIONS:
Device: BabySlide — Application of BabySlide during vacuum-assisted births for perineal protection
  Arms: intervention

SUMMARY:
Visible birth tears are common in vaginal births, especially in vacuum-assisted births. One aim of obstetrical work is to minimize such injuries by an adequate birth management , for example with a proper perineal support. The medical device "BabySlide®" was developed as an auxilliary device for perineal support and already evaluated in a multicenter randomized controlled trial in Schweden in pregnant women during vaginal birth. It could be seen, that the application of the device significantly reduced the rate of vagibal tears and low-grade perineal tearsin the intervention group (with application of the BabySlide®) in contrast to the controlo group (without application of the BabySlide®) by about 10%. In this study, solely 10% of births were ended by vacuum assistance. However, birth tears appear much more often in vacuum-assisted births than in normal spontaneous births. Therefore, the aim of this study is to evaluate the application of the device explicitly in vacuum-assisted births and to investigate if the application should be recommende in vacuum extractions in general in the future.

ELIGIBILITY:
Inclusion Criteria:

* Schwangere Frauen ab 18 Jahren
* Schwangerschaftsalter ab 36+0 SSW bei Geburt
* Einlingsschwangerschaft
* Schädellage des Kindes bei Geburt
* Anstreben einer Vaginalgeburt am USZ
* Geburtsbeendigung per Vakuumextraktion (Saugglocke)
* Schriftliche Einwilligung der teilnehmenden Person nach erfolgter Aufklärung (ausreichende Deutsch- bzw. Englischkenntnisse)

Exclusion Criteria:

* - Geburtsbeendigung per Spontangeburt, Forcepsextraktion (Zange) oder Sectio caesarea (Kaiserschnitt)
* Maternale Erkrankung des Bindegewebes (z.B. Kollagenosen)
* Äusserliche fetale Fehlbildungen, die den Geburtsablauf und die Grössenverhältnisse von Kind zu Geburtskanal verändern
* Intrauteriner Fruchttod des Kindes
* Vaginale, perineale und/oder vulväre Voroperationen (ausser Naht von Geburtsverletzungen)
* St.n. Beckenboden-Operation oder Inkontinenz-Operation
* St.n. Infibulation
* Anwendung des EPI-NO® Dammtrainers während der Schwangerschaft
* Bekannte Allergien gegenüber einem der Inhaltsstoffe des BabySlide®

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
rate of vaginal tears | at day of birth
  assessment of the rate of vaginal tears in the posterior compartment by inspection
rate of low-grade perineal tears | at day of birth
  assessment of the rate of low-grade perineal tears by inspection

SECONDARY OUTCOMES:
rate of high-grade perineal tears | at day of birth
  assessment of the rate of high-grade perineal tears by inspection
Maternal adverse effects | within 1-4 days after birth
  assessment of maternal adverse effects of the BabySlide by medical staff
Fetal adverse effects | within 1-4 days after birth
  assessment of fetal adverse effects of the BabySlide by medical staff
Maternal comfort with the BabySlide | within 1-4 days after birth
  Assessment of maternal comfort with the BabySlide by a questionnaire
User abilitiy | directly after the procedure
  Assessment of the user ability of the BabySlide by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kimmich, Dr., Principal Investigator — University Hospital Zurich, Department od Obstetrics
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided